CLINICAL TRIAL: NCT02092662
Title: Objective Assessment of Upper Extremity Functioning of Stroke Patients Before and After Rehabilitation
Acronym: AssStrFunc
Status: Completed | Type: Observational
Sponsor: Carmeli Eli (Other)
Responsible Party: Sponsor-Investigator, Carmeli Eli, Professor, University of Haifa
Organization: University of Haifa (Other)
Other Study IDs: UHai920130001
Record Dates: First submitted 2014-03-12; First posted 2014-03-20 (Estimated); Results first posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Stroke: Stroke patients at the subacute phase
  Interventions: Other: stroke
- Healthy controls: healthy age-matched voluntiers
  Interventions: Other: Healthy controls

INTERVENTIONS:
Other: stroke — task-oriented therapy: physical and occupational therapy emphasizing integration of the patients needs, environment and context
  Groups: Stroke
Other: Healthy controls — no treatment
  Groups: Healthy controls

SUMMARY:
The purpose of this study is to evaluate by objective measures the improvement in upper extremity functioning, as reflection of motor learning, in stroke patients in the sub acute phase. The investigators hypothesize that the improvements in daily functioning are partially due to compensation strategies and partially due to motor learning.

DETAILED DESCRIPTION:
Background: Most stroke patients continue to suffer from upper extremity motor deficiencies even after prolonged and intense rehabilitation in hospital. Even though guidelines and other studies recommend to apply a rehabilitation programs as patient reception. As opposed to that there is a scarce evidence for the efficacy of the rehabilitation.

Objectives: To evaluate by objective measures the improvement in motor performance of the upper extremity of stroke patients in the sub acute period. Secondary objective is to describe the correlation between proximal and distal motor deficiencies of the upper extremity.

Hypothesis: Patients will show better hand performance at the end of hospitalization. Part of it can be attributed to the rehabilitation and part to a spontaneous recovery. Correlation will be found for proximal and distal upper extremity motor deficiencies.

Methods:

Trial began only after the IRB research approval. All treatment sessions will implemented by the physical and occupational staff of the hospital. Assessments for the measures will be carry out by a certified physical therapist which is coinvestigator. The coinvestigator collect the raw data for analysis in Excel and than in SPSS.

20 stroke patients who meet the inclusion criteria will participate in the study, after signing an informed consent.Patients will undergo the first assessment of all measures, e.g: motor abilities by Fugl-Meyer test, handwriting kinematic and kinetic measures and surface electromyography for measurement of muscle synergy.Patients will be treated by standard rehabilitation of physical and occupational therapy for a period of 3-4 weeks. Before discharge from hospital patients will undergo another assessment of all measures, in order to evaluate the progression in their upper limb motor abilities from reception. Part of the patients will be assessed again two to three weeks after discharge as follow up.

Outcome Measures: upper limb Fugl-Meyer assessment, handwriting Air-time, pressure and velocity, EMG (i.e., muscle onset, muscle amplitude, muscle co-activation ratio).

Statistical analysis: ANOVA analysis will be used to measure time effect. Correlation between measures will be measured by Pearson's correlation. Sample size (n=20) was calculated based on 5 points improvement in Fugl-Meyer test as minimal significant change with power of 0.8 and p-level under 0.05 for significance.

Key words: Stroke, Muscle synergy, Handwriting, Fugl-Meyer

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of cerebral stroke with upper extremity hemiparesis
* Ability to understand simple orders

Exclusion Criteria:

* Other orthopedic pathology
* Apraxia
* Bilateral Paresis
* Other neurologic pathology
* sensory aphasia

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort will be selected from Fliman Rehabilitation Geriatric Center. Healthy subjects, age and gender-matched will be served as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel Markovich, MD, Principal Investigator — Fliman Geriatric Rehabilitation Center; Sharon Israely, MSc., Study Director — University of Haifa; Eli Carmeli, PhD., Study Chair — University of Hifa
Locations (1):
- Fliman Geriatric Rehabilitation Center, Haifa, Israel, Israel

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients After a Stroke: Patients who admitted to the hospital for rehabilitation after a stroke
- Control: Healthy voluntiers
Period: Overall Study
Arm/Group | Patients After a Stroke | Control
Started | 38 | 19
Recruited | 38 | 19
Completed | 25 | 19
Not Completed | 13 | 0
Not completed — Lost to Follow-up | 13 | 0

BASELINE CHARACTERISTICS:
Population: groups were matched by age (p>0.1)
Groups:
- Study: patients after a stroke
- Control: healthy volunteers
- Total: Total of all reporting groups
Arm/Group | Study | Control | Total
Number analyzed (Participants) | 38 | 19 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 34 | 16 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.15 (8.69) | 71 (10.58) | 74 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 25 | 8 | 33
Region of Enrollment [Number; unit: participants]
  Israel | 38 | 19 | 57

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Assessment.
Description: zero to 66 points scale, measuring the impairment level of the upper extremity. Zero indicates a high level of impairment or minimum hand motor function, while 66 points indicates an increased motor function which is similar to normal upper extremity function.
Time Frame: T1 at the beginning of the hospital stay and folloew up at T2 one month later.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Study Group (T1): Patients after a stroke
- Control: Healthy age-matched
Arm/Group | Study Group (T1) | Control
Number analyzed (Participants) | 38 | 19
units on a scale
  Fugl-Meyer assessment score (T1) | 38.32 (13.77) | NA (NA) — Fugl-Meyer assessment intended to evaluate the motor impairment level after a storle, so it was evaluated only in the study group.
  Fugl-Meyer assessment score (T2) | 47.6 (11.06) | NA (NA) — please see T1 assessment above

2. Secondary Outcome: Muscle Co-activation Index.
Description: Assessed by surface electromyography device. Indicate for the level by which muscles contract at the same time and amplitude. It will be calculated in percentage from 100%, as 100% indicate for complete co-activation between a pair of muscles.
Time Frame: T1 at the beginning of the hospital stay and folloew up at T2 one month later.
Reporting Status: Not Posted

3. Secondary Outcome: Handwriting Velocity
Description: Assessed by electronic tablet with specific software called ComPET. Patient make writing tasks. The velocity of his writing is measured and pass from the tablet to the computer to be processed by the software.
Time Frame: T1 at the beginning of the hospital stay and follow up at T2 one month later.
Reporting Status: Not Posted

4. Primary Outcome: Muscle Onset Time.
Description: Assessed by surface electromyography device. The time period it takes the muscle to be activated and contract from a voice prompting is measured. Shorter time onset probably charcterized healthy people compared to patients after a stroke.
Time Frame: the study group was assessed T1 at the beginning of the hospital stay and follow up at T2 one month later. The control group assessed for the the time onset and compared to the study group at T1
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Healthy Controls: healthy age-matched voluntiers
  Healthy controls: no treatment
  Deltoid onset time 0.79 sec
Arm/Group | Stroke | Healthy Controls
Number analyzed (Participants) | 38 | 19
seconds
  Deltoid T1 assessment | 1.33 (0.7) | 0.79 (0.32)
  Deltoid T2 assessment | 0.9 (0.38) | NA (NA) — The control group used to compare the impairment level of stroke patients to healthy aged matched people, so it was not necessary to make to evaluations for the control group.
  Trapezius T1 assessment | 1.09 (0.46) | 0.79 (0.3)
  Trapezius T2 assessment | 0.8 (0.36) | NA (NA) — The same as above
  Biceps T1 assessment | 1.37 (0.7) | 0.79 (0.31)
  Biceps T2 assessment | 0.82 (0.4) | NA (NA) — The same as above
  TricepsT1 assessment | 0.91 (0.81) | 0.72 (0.64)
  Triceps T2 assessment | 1.12 (0.74) | NA (NA) — The same as above

5. Secondary Outcome: % Maximum Voluntary Contraction.
Description: T1 at the beginning of the hospital stay and folloew up at T2 one month later.
Time Frame: The outcome will be measured twice. First at the beginning of the hospital stay and again at the end of the hospital stay, that is 4 weeks on average.
Reporting Status: Not Posted

6. Secondary Outcome: Handwriting Pressure.
Description: Assessed by electronic tablet with specific software called ComPET. Patient make writing tasks, and the pressure exerted with the pen on the tablet is recorded. The data from the tablet passed to the computer to be processed by the software.
Time Frame: T1 at the beginning of the hospital stay and folloew up at T2 one mont...
Reporting Status: Not Posted

7. Secondary Outcome: Handwriting Off-paper Time.
Description: Assessed by electronic tablet with specific software called ComPET. Patient make writing tasks. The time the pen is on air is measured. The data from the tablet passed to the computer to be processed by the software.
Time Frame: T1 at the beginning of the hospital stay and folloew up at T2 one mont...
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: THere were no adverse events in the study
Arm/Group | Study
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No